CLINICAL TRIAL: NCT03120143
Title: Effect of Small-sided Team Sport Training and Protein Intake on Muscle Mass, Physical Function and Markers of Health in Older Untrained Adults
Brief Title: Small-sided Ball Game Training and Protein Intake in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Copenhagen Municipality, Denmark (Other Government); Nestlé Institute of Health Sciences (Unknown)
Responsible Party: Principal Investigator, Jacob Vorup, Principal Investigator, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-15002409
Record Dates: First submitted 2017-04-10; First posted 2017-04-19 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Physical Activity
Keywords: Small-sided ball games; Aging; Muscle mass; Health; Training; Protein intake; Physical function; Physiological adaptations
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Team sport and high protein group (Experimental): This group participated in team sport based small-sided ball games with supplementation of a drink with a high content of protein after the training sessions
  Interventions: Other: Small-sided ball game training with high protein intake
- Team sport and low protein group (Experimental): This group participated in team sport based small-sided ball games with supplementation of a drink low in protein content after the training sessions
  Interventions: Other: Small-sided ball game training with low protein intake
- Control group (No Intervention): This group continued their usual life style without intervention

INTERVENTIONS:
Other: Small-sided ball game training with high protein intake — In the present study, small-sided ball game training consists of repeated intervals of floorball and cone ball training on small areas and 3-4 participants on each team. The supplementation high in protein consists of 18 g protein consumed immediately after and 3 h post exercise
  Arms: Team sport and high protein group
Other: Small-sided ball game training with low protein intake — n the present study, small-sided ball game training consists of repeated intervals of floorball and cone ball training on small areas and 3-4 participants on each team. The supplementation low in protein consists of 3 g protein consumed immediately after and 3 h post exercise.
  Arms: Team sport and low protein group

SUMMARY:
The effect of small-sided team sport training and protein intake on muscle mass, physical function, and adaptations important for health in untrained older adults was examined. Forty-eight untrained older (72±6 years) men and women were divided into either a team sport group ingesting a drink high in protein (18 g) immediately and 3 h after each training session (TS-HP, n=13), a team sport group ingesting an isocaloric drink with low protein content (3 g; TS-LP, n=18), and a control group continuing their normal activities (CON, n=17).

ELIGIBILITY:
Inclusion Criteria:

* adults aged 65 years or older

Exclusion Criteria:

* severe cardiovascular or neurological disease and participation in regular intense exercise training or sports

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Muscle mass | 12 weeks
  Lean body mass in kg determined by DXA scanning

SECONDARY OUTCOMES:
Physical function | 12 weeks
  Sit to stand performance (repetitions in 30 s)

REFERENCES:
- [Derived] Vorup J, Pedersen MT, Brahe LK, Melcher PS, Alstrom JM, Bangsbo J. Effect of small-sided team sport training and protein intake on muscle mass, physical function and markers of health in older untrained adults: A randomized trial. PLoS One. 2017 Oct 10;12(10):e0186202. doi: 10.1371/journal.pone.0186202. eCollection 2017. PMID 29016675